CLINICAL TRIAL: NCT03878017
Title: Feasibility of a Novel Method of Axilla Staging by Using Ultrasound Visible Clips to Mark the Involved Axillary Lymph Nodes Before Neoadjuvant Chemotherapy in Breast Cancer Patients
Brief Title: A Novel Method of Clipped Axillary Lymph Node Localization Post Neoadjuvant Chemotherapy in Breast Cancer Patients .
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Lim Geok Hoon, Senior consultant, KK Women's and Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/2037
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- skin marking of clipped axillary LN (Experimental): all eligible patients underwent skin marking of their clipped axillary LN post neoadjuvant chemotherapy to determine the retrieval rate of the clipped nodes
  Interventions: Procedure: skin marking of clip axillary lymph node for localisation

INTERVENTIONS:
Procedure: skin marking of clip axillary lymph node for localisation — to determine the feasibility of skin marking to localize clipped ln

SUMMARY:
to determine the feasibility of a novel technique of localization of clipped LN post neoadjuvant chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patients with involved axillary LN <3,
* going for neoadjuvant chemotherapy

Exclusion Criteria:

-stage 4 breast cancer patients

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
retrieval rates of the clipped node using this novel technique | at an average of a year

CONTACTS AND LOCATIONS:
Overall Officials: Geok H Lim, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Lim GH, Al Shukairi AM, Lee YS, Teo SY, Yan Z, Tan QT, Gudi M, Ng RP, Wong FY. Targeted axillary dissection in breast cancer patients with metastatic nodal disease: a prospective study on localization techniques and oncological outcomes. Gland Surg. 2025 Aug 31;14(8):1529-1538. doi: 10.21037/gs-2025-166. Epub 2025 Aug 20. PMID 40948928